CLINICAL TRIAL: NCT01254435
Title: Does Patient Position During Extubation at Colonoscopy Influence the Quality of Mucosal Visualisation?
Brief Title: Positioning During Colonoscopy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Steven Brown, Sheffield Teaching Hospitals NHS Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STH14709
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-03

CONDITIONS: Colonic Polyps
Keywords: Colonoscopy; Positioning in colonoscopy; Quality control
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'Free' positioning withdrawal (Active Comparator): Withdrawal of the colonoscope with the patient positioned at the discretion of the endoscopist
  Interventions: Procedure: Colonoscopy
- 'Fixed' position withdrawal (Experimental): Patient positioned in the left lateral position to visualise the caecum, ascending colon and hepatic flexure; supine to visualise the transverse colon; and in the right lateral position to visualise the splenic flexure, descending colon and the sigmoid colon
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Recording of colonoscopic extubation

SUMMARY:
Colonoscopy is the gold standard investigation in the screening of colorectal neoplasms. The investigators hypothesise that visualisation of the colonic mucosa on extubation may be improved by changing patient position as follows: left lateral position for the right colon, supine for the transverse colon and right lateral position for the left colon(fixed positioning). The investigators aim to validate our hypothesis by performing a randomised control study, comparing mucosal visualisation in patients placed in the 'routine' positions at the discretion of the endoscopist with visualisation in those placed in the above described positions. The hypothesis is that fixed positioning confers an advantage.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring colonoscopy

Exclusion Criteria:

* Polyp surveillance
* Cancer surveillance
* Infirmity
* Pregnancy
* Colectomy
* Poor tolerance
* Failed colonoscopy
* Poor bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Mucosal visualisation | 3 months
  Made by video assessment of colonoscopic withdrawal
Luminal distension

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Brown, MD FRCS, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Stuart Riley, FRCP, Study Director — Sheffield Teaching Hospitals NHS Foundation Trust; Wal Baraza, MRCS, Study Chair — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom